CLINICAL TRIAL: NCT00703586
Title: A Two-Arm, Single Site, Proof of Concept Study of the Antiviral and Immunological Effects of Intensification of Suppressive Antiretroviral Therapy With Maraviroc, a CCR5 Antagonist (ADARC 2007-02)
Brief Title: Study of the Antiviral and Immunological Effects of Intensification of Suppressive Antiretroviral Therapy With Maraviroc
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rockefeller University (Other)
Collaborators: Aaron Diamond AIDS Research Center (Other); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MMA-0612
Record Dates: First submitted 2008-06-19; First posted 2008-06-23 (Estimated); Last update posted 2012-10-23 (Estimated); Status verified 2012-10

CONDITIONS: HIV Infections
Keywords: Maraviroc; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): ARM A:
  Intensification with maraviroc for 24 weeks at one of the following doses:
  * 150 mg orally BID when coadministered with a ritonavir-boosted protease inhibitor
  * 600 mg orally BID when coadministered with efavirenz or nevirapine
  Interventions: Drug: Maraviroc
- 2 (Active Comparator): ARM B
  Intensification with an additional NRTI for 12 weeks then cross over to maraviroc intensification for an additional 12 weeks as above:
  * Addition of abacavir 600 mg orally once daily to a tenofovir containing regimen for 12 weeks then replacing the abacavir with maraviroc
  * Addition of an alternate FDA approved NRTI [such as zidovudine (AZT) or didanosine (ddi)] at standard oral dosing to a tenofovir containing regimen for 12 weeks (if the participant declines abacavir therapy) then replacing the alternate NRTI with maraviroc.
  Interventions: Drug: Maraviroc

INTERVENTIONS:
Drug: Maraviroc — ARM A:
  Addition of maraviroc to baseline ARV medications for 24 weeks at one of the following doses:
  * 150 mg orally BID when coadministered with a ritonavir-boosted protease inhibitor
  * 600 mg orally BID when coadministered with efavirenz or nevirapine
  ARM B:
  Addition of an additional NRTI to baseline ARV medications for 12 weeks then cross over to maraviroc intensification for an additional 12 weeks as above:
  * Addition of abacavir 600 mg orally once daily to a tenofovir containing regimen for 12 weeks then replacing the abacavir with maraviroc.
  * Addition of an alternate FDA approved NRTI [such as zidovudine (AZT) or didanosine (ddi)] at standard oral dosing to a tenofir containing regimen for 12 weeks (if the participant declines abacavir therapy) then replacing the alternate NRTI with maraviroc.
  * Addition of tenofovir 300 mg daily to an abacavir containing regimen for 12 weeks then replacing the tenofovir with maraviroc.

SUMMARY:
Hypothesis: Intensification of current ARV regimens with maraviroc will result in more complete suppression of viral replication, particularly in the gastrointestinal mucosa with resultant reduction in markers of immune activation and improved GI immune reconstitution.

DETAILED DESCRIPTION:
* DURATION: Subjects will participate for a minimum of 28 weeks.
* SAMPLE SIZE: 18 subjects randomized 2:1 continued ARVs plus maraviroc versus continued ARVs plus additional ARV to be determined based on baseline ARV regimen.
* REGIMEN: At entry, subjects will be randomized to one of the following in a 2:1 ratio:

ARM A:

Intensification with maraviroc for 24 weeks at one of the following doses:

* 150 mg orally BID when coadministered with a ritonavir-boosted protease inhibitor
* 600 mg orally BID when coadministered with efavirenz or nevirapine

ARM B

Intensification with an additional NRTI for 12 weeks then cross over to maraviroc intensification for an additional 12 weeks as above:

* Addition of abacavir 600 mg orally once daily to a tenofovir containing regimen for 12 weeks then replacing the abacavir with maraviroc
* Addition of an alternate FDA approved NRTI [such as zidovudine (AZT) or didanosine (ddi)] at standard oral dosing to a tenofovir containing regimen for 12 weeks (if the participant declines abacavir therapy) then replacing the alternate NRTI with maraviroc.

The objectives of this study are:

To determine whether intensification of current ARV regimens with maraviroc will result in more complete suppression of viral replication and improved immune reconstitution in GI mucosal lymphoid compartment based on:

* Reduction in normalized levels of CD4+MMC HIV-1 RNA as determined by PCR pre- and post- intensification at week 12 in Arm A versus Arm B.
* Reduction in normalized levels of CD4+ mucosal mononuclear cell (MMC) HIV-1 RNA at week 12 compared to baseline in Arm A.
* Reduction in %CD4+MMC HIV-1 RNA positive as determined by PCR pre- and post- intensification between Arm A and Arm B as well as week 12 and 24 post maraviroc intensification.
* Levels of CD4+ T cells in GALT (% by flow and absolute #s by immunohistochemistry).
* Phenotype of cells in GALT by flow (memory, naive, R5, X4, dual expressing).
* Levels of activation of CD4 and CD8 in PB and GALT using HLA DR and CD 38.

ELIGIBILITY:
Inclusion Criteria:

* Documented treatment with combination antiviral therapy (ARV) during acute and early HIV-1 infection defined as:

  * Negative ELISA/Western Blot or indeterminate Western Blot in the presence of HIV-1 RNA>5,000 copies/ml
  * Positive HIV-1 serology with a detuned ELISA O.D. value below 1.0
  * A documented negative serology within 180 days of screening and a positive HIV-1 serology at screening
* Treatment for at least one year with ARVs
* Plasma HIV-1 RNA levels below detection for at least 6 months
* CCR5 tropic virus pretreatment using the Monogram assay
* GI biopsy at study entry
* Agree to subsequent GI biopsy at 12 and 24 weeks
* Laboratory values obtained within 45 days prior to study entry.

  * Absolute neutrophil count (ANC) ≥500/mm³
  * Hemoglobin ≥9.0 g/dL
  * Platelet count ≥80,000/mm³
  * AST (SGOT), ALT (SGPT), and alkaline phosphatase < 5.0 x ULN
  * Total bilirubin ≤ 2.5 X ULN if not on atazanavir containing regimen
  * PT/PTT within 1.5 control
  * Calculated creatinine clearance ≥60 mL/min as estimated by the Cockcroft Gault equation:
  * For men, (140 - age in years) x (body weight in kg) / (serum creatinine in mg/dL x 72) = CrCl (mL/min)
  * For women, multiply the result by 0.85 = CrCl (mL/min) NOTE: A program to assist in calculations is available on the DMC web site at: http://www.fstrf.org/ACTG/ccc.html
* For women of reproductive potential, negative serum or urine pregnancy test within 48 hours prior to initiating study medications unless otherwise specified by product labeling.
* Female candidates of reproductive potential is defined as girls who have reached menarche or women who have not been post-menopausal for at least 24 consecutive months (i.e., who have had menses within the preceding 24 months) or have not undergone surgical sterilization (e.g., hysterectomy, or bilateral oophorectomy, or bilateral tubal ligation).
* Contraception requirements:

  * Female candidates of reproductive potential, who are participating in sexual activity that could lead to pregnancy, must agree that they will use at least one reliable method of contraception while receiving the protocol-specified drugs and for 6 weeks after stopping the medications.
  * Male Candidates: If you are a heterosexual male, you and your sexual partner must agree to use acceptable methods of birth control during the entire study. Acceptable methods of birth control include intrauterine device (IUD), diaphragm with spermicide,condoms or not having sex. Oral contraceptives alone are not an acceptable method of birth control.
* Men and women age ≥18 years.
* Participants must be HLA-B5701 negative if not taking abacavir as part of their regimen.
* Ability and willingness of subject to give written informed consent.

Exclusion Criteria:

* Currently breast-feeding.
* Use of immunomodulators (e.g., interleukins, interferons, cyclosporine), HIV vaccine, systemic cytotoxic chemotherapy, or investigational therapy within 30 days prior to study entry. NOTE: Subjects receiving stable physiologic glucocorticoid doses, defined as prednisone ≤ 10 mg/day, will not be excluded.
* Known allergy/sensitivity to study drugs or their formulations.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Serious illness requiring systemic treatment and/or hospitalization until candidate either completes therapy or is clinically stable on therapy, in the opinion of the site investigator, for at least 7 days prior to study entry.
* Pretreatment viral population that is either dual mixed tropic or X4 tropic using the Monogram assay
* Current imprisonment or involuntary incarceration in a medical facility for psychiatric or physical (e.g., infectious disease) illness.
* Any other clinical conditions or prior therapy that, in the opinion of the investigator, would make the subject unsuitable for the study or unable to comply with the requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
MMC HIV RNA | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Martin Markowitz, MD, Principal Investigator — Rockefeller University
Locations (1):
- Rockefeller University Hospital, New York, New York, United States